CLINICAL TRIAL: NCT02728713
Title: Effect of Osteopathic Cranial Manipulative Medicine on Visual Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Osteopathic Heritage Foundations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HPD-OST07220201
Record Dates: First submitted 2014-04-03; First posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Visual Function
Keywords: Cranial manipulation; Visual function

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Cranial manipulation (Experimental): Assessment for cranial strain patterns, followed by indirect cranial manipulation to treat dysfunctions found on assessment, followed by reassessment.
  Repeated for a total of eight visits no less than one week apart.
  Interventions: Procedure: Cranial Manipulation
- Sham/placebo (Sham Comparator): Assessment for cranial strain patterns, followed a laying on of hands, followed by reassessment. Repeated for a total of eight visits no less than one week apart.
  Interventions: Procedure: Sham/Placebo

INTERVENTIONS:
Procedure: Cranial Manipulation — Performed by exaggerating the motion asymmetry with a minimum of pressure (a few ounces) and holding the position until the motion becomes symmetrical.
  Other Names: Osteopathy in the Cranial Field; Osteopathic Cranial Manipulative Medicine
  Arms: Cranial manipulation
Procedure: Sham/Placebo — A laying on of hands with no actual treatment being performed.
  Arms: Sham/placebo

SUMMARY:
The purpose of this study is to determine if there is a measurable change in visual function as a direct result of the application of osteopathic cranial manipulative medicine. The study will also attempt to determine whether any changes noted remain after withdrawal of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* free of active ocular or systemic disease
* refractive error between six diopters of myopia and five diopters of hyperopia with regular astigmatism of any amount
* normal best-corrected visual acuity at 20/40 or better
* normal amplitude of accommodation
* willing to undergo osteopathic cranial manipulative medicine

Exclusion Criteria:

* pregnancy
* history of previous closed head trauma or brain injury
* prior cranial manipulative treatment/craniosacral therapy
* students from the Nova Southeastern University Colleges of Osteopathic Medicine and Optometry

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2003-08; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Distance Visual Acuity | Weekly for 16 weeks
  Measurement of visual acuity in each eye by number of letters read correctly on ETDRS chart.
Accommodative System Testing | Weekly for 16 weeks
  Accommodative amplitude testing using a Donder push-up card.
Local Stereoacuity Testing | Weekly for 16 weeks
  Measured by Random Dot E test.
Pupillary Size Testing | Weekly for 16 weeks
  Measurement of pupil size (each eye) in bright and dim light.
Vergence System Testing | Weekly for 16 weeks
  Assessed by Cover Test with Prism Neutralization and Near Point of Convergence

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sandhouse, D.O., M.S., Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University Davie Health Center, Fort Lauderdale, Florida, United States

REFERENCES:
- [Derived] Sandhouse ME, Shechtman D, Fecho G, Timoshkin EM. Effect of Osteopathic Cranial Manipulative Medicine on Visual Function. J Am Osteopath Assoc. 2016 Nov 1;116(11):706-714. doi: 10.7556/jaoa.2016.141. PMID 27802556